CLINICAL TRIAL: NCT06516250
Title: GEMAS Proyect. Gamification in Nursing and Medicine for Simulation Learning.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Munir Mohamed Mimun, Principal investigator, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GEMASMMM2024
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Serious game; Simulation; Gamification; Knowledge; Learning methodologies; Urgency; Emergency
MeSH Terms: conditions — Behavior; Emergencies

STUDY DESIGN:
Intervention Model Description: Students enrolled in 5th and 6th year medicine or 3rd and 4th year nursing degree programs. They can be from various faculties.
  Residents in training in medicine or nursing, from various years of residency and specialties.
Who Masked: Outcomes Assessor
Masking Description: Once the data is obtained, it will be sent to the results analysts who will also not know the authorship of the data obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with serious game (Experimental): The participants will recived the same theoretical master classes and they will use the serious game for a series of hours and will be able to learn using this new teaching methodology, whether on a computer or mobile.
  Interventions: Other: Virtual serious game GEMAS
- Group traditional methods of learning (No Intervention): They will not be able to use the application, its teaching method will be based on theoretical master classes.

INTERVENTIONS:
Other: Virtual serious game GEMAS — Implement and evaluate a virtual serious game designed to improve the learning and retention of clinical knowledge in medicine and nursing students and residents through the simulation of clinical cases in a hospital emergency environment.
  Arms: Group with serious game

SUMMARY:
The GEMAS project is based on the creation of a virtual serious game in which, by carrying out clinical cases that simulate real environments and episodes of a hospital emergency service, the aim is to improve and reinforce the knowledge of the participants with the use of a new learning methodology.

The mapping and creation of several scenarios within the program is carried out, the creation of different characters, both main and secondary, patients and hospital environment, each of them with their graphic representation, characteristics and individual personality.

After obtaining the program, which can be used on both computer and mobile platforms, the virtual serious-game will be evaluated with the levels of the Kirkpatrick model to be used as a new learning tool. The degree of satisfaction and usability will be evaluated at the first level, the degree of knowledge acquisition by the participant himself and in comparison with traditional methodologies at the second level, the changes in behavior and transfer of the knowledge learned to the professional field in the third level, and the possibility of knowing the effectiveness of the application for the system will be evaluated. The virtual serious game will allow you to select between the nursing or medicine modality, allowing a greater number of cases to be developed and at the same time, for both stories to be related, so that interdisciplinarity remains intrinsically rooted in the game. The creation of this application will create dynamic learning that will allow greater user satisfaction while learning and a greater degree of knowledge acquisition with respect to traditional methods, ultimately producing changes in work behavior that are favorable for the performance of their profession. .

DETAILED DESCRIPTION:
Specific Objective 1

The design of the application will be carried out using the RPG Maker MV program, an online purchase programming tool that grants the buyer intellectual property and commercialization rights. After acquiring the program, a hospital environment will be created, in this case, an Emergency Medical System, creating different characters including patients, family members, doctors, nurses, and administrative staff. The stories will be divided into two for gameplay, depending on whether the player chooses to be a nurse or a doctor. Consequently, the stories are different, and the characters represent a series of cases and varying complexity, adapted to the decision of which profession to pursue in the game. The characters will be created using the Midjourney™ web application as sketches, which will then undergo multiple image changes with GIMP 2.10, Paint, and PowerPoint until the desired images of the different characters are achieved.

In the content of the virtual serious game, two stories will be created with the intention of learning about various common deficits or errors made by novice doctors and nurses.

To design the content, an expert group will be formed, requesting the participation of professionals with extensive experience in the field of medical emergencies and nursing with an interdisciplinary vision, who wish to participate in the creation of case content.

Specific Objective 2

To evaluate the degree of satisfaction and usability of the virtual serious game, surveys or questionnaires will be used. The degree of usability will be measured using the SUS (System Usability Scale), which aims to assess navigation, interface design, and accessibility. This scale, created in 1986 by John Brooke, is widely validated for measuring the usability of systems and products, including software, hardware, mobile applications, and other interactive systems. It is based on responses to 10 items rated on a 4-point Likert scale (from strongly disagree to strongly agree).

Direct observation of the game functioning will also provide feedback on programming, image, and development errors in the application, allowing us to make the necessary modifications.

To assess the degree of satisfaction, the 9-question Kirkpatrick model questionnaire will be used, presenting questions with Likert scale ratings and open-ended questions. Additional questions from the Questionnaire for User Interaction Satisfaction (QUIS), a widely validated scale used to evaluate user satisfaction with interaction systems, including software and educational applications, will be added. This will complement the Kirkpatrick scale due to the lack of questions evaluating interactions with software and computer systems. The QUIS was developed at the Human-Computer Interaction Lab at the University of Maryland and has been validated through multiple academic studies and practical applications. This scale traditionally scores from 1-very dissatisfied to 9-very satisfied, evaluating various aspects of user satisfaction. The QUIS questions that best address the information we want to obtain from the project will be selected and added to the Kirkpatrick level 1 model questions.

Specific Objective 3

To evaluate the degree of clinical knowledge acquired, a knowledge questionnaire will be designed in conjunction with a consensus of experts using the Delphi method. For the creation of the questionnaire, a literature review will be conducted to establish that there is currently no agreement among researchers on using a scale that measures the knowledge we want to evaluate and reinforce in the students. Therefore, the question "How can I evaluate the knowledge of virtual serious game participants before and after its use to know the degree of learning acquired?" will be posed.

Once the absence of such a scale is identified, a group will be constituted to coordinate the process, comprising the thesis directors and the doctoral candidate. The functions will include creating a group of experts in emergency medicine and nursing to contribute their knowledge and involvement in improving knowledge for our project. A study and approval of the expert list will be conducted, the questionnaire will be developed, expert participation will be encouraged, responses from the rounds will be analyzed, subsequent questionnaires or questions will be prepared and feedback provided, and the process will be supervised, proposing and taking corrective measures if necessary, and ultimately interpreting the results. Feedback will serve as the link between the experts and the coordinators, allowing information flow and improving the final product quality.

Specific Objective 4

During the beginning of residency, both nurses and doctors are instructed in preparatory classes before starting their shifts and rotations in the Emergency Department. Two groups will be selected: an intervention group that will use the virtual serious game after the lectures given at the center, and a control group that will follow the traditional lecture method for knowledge acquisition.

The intervention group will be allowed to enjoy the virtual serious game for the hours needed to advance through the difficulty levels until completing 100% of the virtual serious game. Subsequently, as indicated in objective 3, a post-test will be administered, collecting responses on the knowledge that the virtual serious game and the emergency lectures are expected to cover.

In the control group, after attending lectures that cover the topics addressed by the virtual serious game, the same post-test will be administered. This way, we can determine whether the use of the virtual serious game is favorable for clinical knowledge acquisition by producing statistically significant results compared to the control group.

Participant selection for both groups will follow a series of steps:

Participant acceptance according to inclusion and exclusion criteria and their willingness to participate in the study.

Sample stratification, separating doctors and nurses, and those who have previously worked or are in their second residency from the more novice participants.

Randomization of participants into the control and intervention groups using randomization software or a traditional random number table method.

Assignment by a third person, avoiding, as much as possible, the ability of the person assigning participants to identify them. This would be achieved by using identification codes instead of participant names.

Specific Objective 5

To evaluate the application of the virtual serious game for clinical case simulation as a preparation tool for the Objective Structured Clinical Examination (OSCE), a methodology similar to that described in objective 4 will be used. However, in this case, samples will be obtained from medical and nursing students, who will consent to participate in the study and to share their OSCE scores for evaluation.

The selection of intervention and control groups will be made by selecting users who want to participate in the study before the OSCE. Those students who meet the inclusion and exclusion criteria will be selected through stratified (by faculty and geographic location) and randomized allocation to the intervention and control groups. The selection will be blinded, resulting in two groups:

Intervention group: Will have access to the application on their mobile phone or PC at the teaching center, being able to complete the game before the OSCE.

Control group: Will take the OSCE using traditional learning and knowledge acquisition techniques currently employed at the center.

Once both groups are obtained and the intervention with the virtual serious game tool is completed, OSCE results will be collected to evaluate whether there are statistically significant differences between the intervention and control groups.

Specific Objective 6

Evaluate behavioral changes in professionals using the application. To do this, the 6-question Kirkpatrick model questionnaire will be used to determine if there are changes in participants' habits and if there are limitations to its use or development.

ELIGIBILITY:
Inclusion Criteria:

* Medical and Nursing Students: Students enrolled in undergraduate programs in medicine (5th and 6th year) or nursing (3rd and 4th year). They may be from various faculties.
* MIR and EIR Residents: Residents in training in medicine or nursing, from various years of residency and specialties.
* Geographic Diversity: Participants from different geographic regions or urban areas.
* Cultural and Linguistic Diversity: Participants from diverse cultures and ethnic groups.
* Willingness to Participate: Commitment of participants to actively participate in the study.

Exclusion Criteria:

* Previous Experience in Similar Cases: Participants who have had previous experience in similar clinical cases or who have received specific training related to the content of the game.
* Severe Mental or Physical Health Issues: Participants who have severe mental or physical health issues that may affect their ability to participate in the study or adequately understand the content of the game.
* Conditions Affecting Active Participation: Participants who have conditions that limit their ability to actively participate in the study (states of intoxication, etc.).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of the virtual serious game | one year
  Measured using the 9-question Kirkpatrick model survey, supplemented with questions from the QUIS (Questionnaire for User Interaction Satisfaction) survey.
  This scale traditionally makes scores from 1- very dissatisfied to 9- very satisfied, evaluating various aspects of user satisfaction such as:
  * Global experience: user's general perception of the system.
  * Screens: design and layout of the screens.
  * Terminology and information system: clarity and appropriateness of the language used.
  * Learning: ease with which users can learn to use the system.
  * System responsiveness: speed and efficiency of system responses.
  * Usability impression: perceived ease of use.
Usability of the virtual serious game | one year
  Usability will be measured with the System Usability Scale (SUS). It is based on providing answers to 10 items that users rate using a 4-point Likert scale (not at all agree 1, to completely agree 4). The items that are evaluated in this scale are:
  Frequency of Use, Complexity. Ease of Use, Need for Technical Support, Integration of Functionalities, Consistency, Ease of Learning, Cumbersomeness, Confidence and Learning Load.
Clinical knowledge | one year
  Measured using a questionnaire validated by a consensus of experts conducted with the Delphi method, with post-test questions added for calibration of the Kirkpatrick method.
  The answer could be correct, partially correct or wrong. The calibration answer are open answer that would give information to the creators to know the subjetive opinion of the participants.
Transfer and behavior after using the serious game modules | one year
  Evaluated using the 6-question Kirkpatrick model survey. The answers would be open answers to know the opinion of the participants and what kind of problems or facilities they have found during the develop of their activities and use of the knowledge and tools achieved during the programme.

IPD SHARING:
Plan to Share IPD: Undecided